CLINICAL TRIAL: NCT01181583
Title: Efficacy Testing of a Tailored Internet-delivered Cognitive Behaviour Therapy Treatment for Symptoms of Depression and Comorbid Problems
Brief Title: Tailored Internet-delivered Cognitive Behaviour Therapy for Symptoms of Depression and Comorbid Problems
Acronym: TAYLOR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Gerhard Andersson/Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-VR-DEP2009-1
Record Dates: First submitted 2010-08-09; First posted 2010-08-13 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tailored Internet-delivered CBT (Experimental)
  Interventions: Behavioral: Tailored Internet-delivered CBT
- Non-tailored Internet-delivered CBT (Experimental)
  Interventions: Behavioral: Non-tailored Internet-delivered CBT
- Online discussion group (Active Comparator)
  Interventions: Behavioral: Online discussion group

INTERVENTIONS:
Behavioral: Tailored Internet-delivered CBT — This intervention contains 8-10 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are "prescribed following the diagnostic telephone interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.
  Arms: Tailored Internet-delivered CBT
Behavioral: Non-tailored Internet-delivered CBT — Specific text-based self-help for depression, which has previously been tested in three previous randomized trials. Anxiety symptoms will not be covered, but insomnia is included as a module together with advice on health.
  Arms: Non-tailored Internet-delivered CBT
Behavioral: Online discussion group — Participants take part of an online discussion group which are monitored daily. New discussion topics on depression are introduced every week.
  Arms: Online discussion group

SUMMARY:
The overall aim of this study is to develop and test a tailored Internet-delivered psychological treatment for patients with mild to moderate major depression and comorbid anxiety symptoms and compare its efficacy to a non-tailored treatment and to an active control group.

DETAILED DESCRIPTION:
Internet-delivered cognitive behaviour therapy (CBT) has emerged as a promising way to administer evidence-based psychological treatments. Mild to moderate major depression has previously been found to treatable via the Internet, with the provision that minimal therapist guidance is given. However, previous research has not taken the issue of comorbidity into account. It is well known that major depression often is accompanied by anxiety and in addition the symptom profile in major depression may differ substantially. The idea behind the proposed research is to tailor the Internet intervention according to the symptom profile. By used a large set of treatment modules (text-based) we aim to diagnose and then prescribe modules. In a randomized trial we want to compare this procedure (e.g., tailored CBT) with the standard Internet-delivered CBT. We will also include a control group in the form of a supervised online discussion group who will later receive CBT.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder
* 15 or more on MADRS-S

Exclusion Criteria:

* Severe depression (more than 35 on MADRS-S or based on interview)
* Severe psychiatric condition (e.g. psychosis or bipolar disorder)
* Changed medication during the last three months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | One week before the treatment starts
Beck Depression Inventory (BDI) | Five weeks after treatment started
Beck Depression Inventory (BDI) | At treatment termination (10 weeks)
Beck Depression Inventory (BDI) | 6 month after treatment ended
Beck Depression Inventory (BDI) | 2 years after treatment ended

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | One week before the treatment starts
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | One week before the treatment starts
Quality of Life Inventory (QOLI) | One week before the treatment starts
Beck Anxiety Inventory (BAI) | Five weeks after treatment started
Beck Anxiety Inventory (BAI) | At treatment termination (10 weeks)
Beck Anxiety Inventory (BAI) | 6 month after treatment ended
Beck Anxiety Inventory (BAI) | 2 years after treatment ended
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | Five weeks after treatment started
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | At treatment termination (10 weeks)
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | 6 month after treatment ended
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | 2 years after treatment ended
Quality of Life Inventory (QOLI) | Five weeks after treatment started
Quality of Life Inventory (QOLI) | At treatment termination (10 weeks)
Quality of Life Inventory (QOLI) | 6 month after treatment ended
Quality of Life Inventory (QOLI) | 2 years after treatment ended

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Department of Behavioral Sciences and Learning, Linköping University
Locations (1):
- Linköping University, Department of Behavioral Sciences and Learning, Linköping, Sweden

REFERENCES:
- [Derived] Johansson R, Sjoberg E, Sjogren M, Johnsson E, Carlbring P, Andersson T, Rousseau A, Andersson G. Tailored vs. standardized internet-based cognitive behavior therapy for depression and comorbid symptoms: a randomized controlled trial. PLoS One. 2012;7(5):e36905. doi: 10.1371/journal.pone.0036905. Epub 2012 May 15. PMID 22615841